CLINICAL TRIAL: NCT07046819
Title: A Randomized, Double-Blind, Placebo-Controlled, Flexible Dose Phase 2 Study of Efficacy and Safety of Tirzepatide in Individuals With Alcohol Use Disorder and Metabolic Alcohol-associated Liver Disease
Brief Title: Tirzepatide in MetALD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 10002246; 002246-AA
Record Dates: First submitted 2025-07-01; First posted 2025-07-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-12

CONDITIONS: Metabolic Alcohol-associated Liver Disease; Alcohol Use Disorder
Keywords: BMI; Weight; Alcohol; Metabolism
MeSH Terms: conditions — Alcoholism; Body Weight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator): A 2.5mg, 5mg, and 7.5mg subcutaneous injection will be given once weekly for 12 weeks.
  Interventions: Other: Placebo
- Tirzepatide (Active Comparator): A 2.5mg, 5mg, and 7.5mg subcutaneous injection will be given once weekly for 12 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — A 2.5mg, 5mg, and 7.5mg subcutaneous injection will be given once weekly for 12 weeks.
  Arms: Tirzepatide
Other: Placebo — A 2.5mg, 5mg, and 7.5mg subcutaneous injection will be given once weekly for 12 weeks.
  Arms: Saline

SUMMARY:
Background:

People with alcohol use disorder (AUD) often develop metabolic alcohol-associated liver disease (MetALD). MetALD is a term for the heart, liver, obesity, and other issues that can accompany AUD. MetALD can be fatal. An approved weight management drug (Tirzepatide) may be able to help people with AUD and MetALD control their alcohol intake.

Objective:

To test Tirzepatide in people with AUD and MetALD.

Eligibility:

People aged 21 years and older with AUD and MetALD.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have a test of their heart function. They will have a Fibroscan: This test uses ultrasound to measure how stiff the liver is. They will answer questions about their alcohol drinking, eating habits, and mental health. Participants may opt to have imaging scans of their brain and liver.

These tests will be repeated in a baseline visit. This visit will take up to 6 hours.

Tirzepatide is injected under the skin once a week for 12 weeks. Participants will visit the clinic to receive each injection. Some participants will get a placebo. A placebo is given just like a Tirzepatide injection but contains no medicine. The physical exam and other tests will be repeated during clinic visits. The Fibroscan will be repeated every 2 weeks during the study. Each weekly visit will take up to 3 hours.

All tests will be repeated on the last visit. These tests will include the imaging scans and Fibroscan. Participants will learn about treatment options for AUD; they will be given recommendations on ways to reduce alcohol intake. This visit will take up to 6 hours.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

The GLP-1/GIP receptor dual agonist tirzepatide has been recently shown to reduce HbA1c in adults with Type 2 diabetes, achieve weight reduction in adults with obesity and reduce metabolic dysfunction associated steatohepatitis. In addition, some data suggest beneficial effects on drinking behaviors. This study will evaluate the efficacy and safety of tirzepatide as a novel treatment for alcohol use disorder (AUD) and metabolic alcohol-associated liver disease (MetALD).

We hypothesize that tirzepatide will be well tolerated and safe in this new target population and that tirzepatide will achieve reduction in alcohol use, metabolic improvement and attenuate alcohol-induced liver steatosis.

OBJECTIVES:

Primary Objective:

The primary objective is to assess the efficacy of tirzepatide in individuals with AUD/MetALD.

Secondary/Exploratory Objectives:

Secondary/exploratory objectives are to assess various biomarkers related to alcohol-induced liver damage, inflammation, neuropsychiatric outcomes, drinking behaviors, epigenetic age acceleration, brain metabolites, and safety.

ENDPOINTS:

Primary endpoints:

- co-primary endpoint: metabolic improvement from baseline as measured by percentage reduction of body weight and reduction in liver steatosis from baseline as measured by percentage reduction in Fibroscan controlled attenuation parameter (CAP) score.

Secondary endpoints:

* Reduction in liver steatosis from baseline as measured by MRI spectroscopy
* Reduction in MRI visceral fat from baseline
* Reduction in liver enzymes (ALT, AST, GGT) from baseline
* Reduction in drinking behaviors/cravings from baseline
* Reduction in one WHO risk drinking level

Secondary safety endpoints:

- Safety and tolerability

Exploratory endpoints:

* Effects on biomarkers (i.e. Il-6, FGF21, epigenetic and genetic markers, proteomics, metabolomics)
* Effects on depression and anxiety measures
* Effects on epigenetic age acceleration
* Changes in brain metabolites as measured by MRI spectroscopy
* Changes in resting state functional connectivity

ELIGIBILITY:
* INCLUSION CRITERIA

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age 21 or older
2. Ability to provide written informed consent
3. Females: Negative urine pregnancy test, not currently breastfeeding, agree to abstain or use accepted form of contraception including use of oral contraceptives and an additional barrier method of contraceptive such as condoms; use of an approved IUD or other longacting reversible contraceptive (LARC); have a male sexual partner who is surgically sterilized; or have exclusively female sexual partner(s)
4. Males: Agree to abstain or use accepted form of contraception, such as condoms.
5. Diagnosis of AUD as confirmed by MINI
6. Current alcohol use as assessed via the TLFB (>14 standard drinks per week for males and >7 standard drinks per week for females on average for the last 8 weeks)
7. Liver steatosis as determined by Fibroscan (CAP score >240) at screening
8. BMI >= 25 and <40 kg/m^2
9. metALD as defined by at least one out of 5 criteria at screening:

   1. BMI >= 25 and <40 kg/m^2
   2. Fasting serum glucose >= 5.6mmol/L [100mg/dL] or HbA1c >=5.7%
   3. Blood pressure >=130/85 or specific antihypertensive drug treatment
   4. Plasma triglycerides >=1.70mmol/L [150mg/dL] or lipid lowering treatment
   5. Plasma HDL-cholesterol less than 1.0mmol/L [40mg/dL] or lipid lowering treatment

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Treatment seeking for alcohol use disorder
2. History of a serious hypersensitivity reaction to GLP-1RA/GIPRA
3. Current/past use of GLP-1RA/GIPRA within the last 3 months
4. Clinically significant and/or unstable cardiovascular disease over the past 12 months
5. History of diabetes mellitus or blood hemoglobin A1c (HbA1c) >= 6.5 % at screening
6. Any underlying clinically significant and/or unstable acute or chronic liver disease unrelated to alcohol use at screening, history of cirrhosis, esophageal varices
7. Subjects with platelets count of less than 110,000/ mm^3
8. Alanine aminotransferase or aspartate aminotransferase exceeding 5 times the upper limit of normal levels at screening
9. Bilirubin 2x UNL or Creatinine > 2 mg/dL at screening
10. Patients with coagulopathy defined as INR >1.5, prothrombin time prolonged by > 3s, and/or platelets <75,000 / mm^3 at screening
11. Positive HIV test or positive Hepatitis B surface antigen (HBsAg), and/or positive Hepatitis C antibody (HCV) at screening
12. Chronic renal failure as estimated by glomerular filtration rate (GFR) < 60mL/min/1.73 m^2 at screening
13. History of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
14. History of previous bariatric surgery or transplant surgery
15. Patients with significant hematologic abnormalities, as defined by hemoglobin < 8g/dL and/or white blood count <1500 cells/microL
16. Current or prior history of any clinically significant disease, including, seizure disorder, epilepsy, alcohol related seizures within 12 months of screening, uncontrolled endocrine disease, hemorrhagic stroke, cancer within the past 5 years or any other significant abnormality identified at the time of screening that, in the judgment of the investigator or study clinician, would preclude safe completion of the study
17. Use of any medications that interfere with tirzepatide
18. Use of the following medications with glucose lowering properties in the last 30 days: GLP-1RA, GLP-1RA/GIPRA, insulin, metformin, sulfonylurea, thiazolidinediones, dipeptidyl peptidase-4 inhibitors, sodium-glucose cotransporter-2 inhibitors
19. Use of the following medications: Any medication that requires intramuscular administration injections. Systemic corticosteroids
20. Use of any investigational drugs within 1 month, or five half-lives, whichever is longer, of the study procedures
21. Presence of any current suicidality or a lifetime history of suicide attempt or suicidal ideation within the past year
22. History of serious mental illnesses including psychotic disorders, bipolar disorders, severe anxiety, mood, or trauma-related disorders and other psychiatric conditions which in the opinion of the investigators would impede the patient's participation or compliance in the study
23. History of liver decompensation events such as hepatic encephalopathy or ascites
24. History of severe gastroparesis
25. History of pancreatitis in the last 5 years or if subject has chronic pancreatitis

For optional MRI: a) Presence of ferromagnetic objects in the body that may be adversely affected by or contraindicated for MRI, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report b) Use of MRI- incompatible intrauterine device (IUD).

Individuals who are pregnant or breastfeeding, or with severe hepatic or renal liver impairment will be excluded from this study because there is no clinical data on the safety of tirzepatide in these populations, including the impact on the fetus or infant. To assess pregnancy status, participants who can become pregnant will be required to take a urine pregnancy test and to test negative before administering study drug.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic improvement from baseline as measured by percentage reduction of body weight and reduction in liver steatosis from baseline as measured by percentage reduction in Fibroscan controlled attenuation parameter (CAP) score. | Change from baseline to week 12

SECONDARY OUTCOMES:
Reduction from baseline in - 1) Liver steatosis as measured by MRI spectroscopy, 2) MRI visceral fat, 3) Liver enzymes (ALT, AST, GGT), 4) Drinking behaviors/cravings, 5) WHO risk drinking level | Change from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Falk W Lohoff, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD relevant to publication will be shared.
Supporting Information: SAP
Time Frame: IPD may be available within 12-24 months of publication.
Access Criteria: IPD may be shared via secured email. The principal investigator will review requests based on specific criteria.

REFERENCES:
- [Background] Coskun T, Sloop KW, Loghin C, Alsina-Fernandez J, Urva S, Bokvist KB, Cui X, Briere DA, Cabrera O, Roell WC, Kuchibhotla U, Moyers JS, Benson CT, Gimeno RE, D'Alessio DA, Haupt A. LY3298176, a novel dual GIP and GLP-1 receptor agonist for the treatment of type 2 diabetes mellitus: From discovery to clinical proof of concept. Mol Metab. 2018 Dec;18:3-14. doi: 10.1016/j.molmet.2018.09.009. Epub 2018 Oct 3. PMID 30473097
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002246-AA.html